CLINICAL TRIAL: NCT05682859
Title: Treatment of Chronic Hand Eczema With Oral Roflumilast (HERO) - a Randomized Controlled Trial
Brief Title: Treatment of Chronic Hand Eczema With Oral Roflumilast (HERO)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jacob Pontoppidan Thyssen (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Sponsor-Investigator, Jacob Pontoppidan Thyssen, Professor, MD, DMSc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC-HE-RO; 2022-503011-42-00 (Other: EU trial number)
Record Dates: First submitted 2022-12-16; First posted 2023-01-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Hand Eczema
MeSH Terms: interventions — Roflumilast; Tablets

STUDY DESIGN:
Intervention Model Description: Multicentre, double-blinded, randomized, placebo-controlled, clinical trial with open-label extension
Who Masked: Participant, Investigator
Masking Description: The investigators as well as the participating patients are blinded during the RCTs phase 1 of roflumilast/placebo. No one is blinded in phase 2 because it is an open-label extension.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roflumilast (Active Comparator): 20 of the participating patients are randomized to the active arm where systemic roflumilast 500 microgram tablets are received.
  Interventions: Drug: Roflumilast 500 Mcg Oral Tablet
- Placebo (Placebo Comparator): 20 of the participating patients are randomized to the active arm where systemic placebo tablets are received.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast 500 Mcg Oral Tablet — Randomized to either systemic roflumilast or placebo in phase 1. All participating patients will receive roflumilast in phase 2.
  Other Names: Daxas
  Arms: Roflumilast
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This study is a multicentre, double-blinded, randomized, placebo-controlled, clinical trial with open-label extension.

The purpose and aim of this study is to investigate the efficacy and safety of roflumilast (PDE4-inhibitor) in adult patients with chronic hand eczema (CHE).

Patients will receive 16-week treatment with either roflumilast or placebo tablets. Hereafter, both groups continue in open-label treatment for 12 weeks where both groups will receive treatment with roflumilast.

DETAILED DESCRIPTION:
This study will investigate the efficacy and safety of roflumilast in adult patients with CHE and it is hypothesized that patients treated with oral roflumilast (500 microgram once daily) will experience an improvement in their moderate-to-severe CHE (measured by hand eczema severity index (HECSI)) and alter the skin microbiome. Secondly, it is hypothesized that patients treated with oral roflumilast will experience improved lung function and weight loss.

This study includes two phases:

Phase 1: 20 patients will receive 500 microgram tablet of roflumilast once daily for 16 weeks while 20 patients will receive placebo once daily for 16 weeks.

Phase 2: All 40 patients from phase 1 will receive 500 microgram tablet of roflumilast once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Age ≤ 75 years
* HECSI ≥ 18 (moderate to severe hand eczema)
* IGA-CHE ≥ 3
* Body mass index (BMI) ≥ 20 kg/m2
* Negative pregnancy test (only women of child-bearing potential (see section 2.8))
* Willing to use safe anticonception during entire study and at least 1 week after end of treatment (-5 times plasma half-life of Roflumilast). This only account for women child-bearing potential
* Speaks, understands, and reads danish.

Exclusion Criteria:

* Severe immunological disease, e.g. HIV, systemic lupus, and systemic sclerosis
* Diagnosis of current tuberculosis
* Current viral hepatitis
* History of heart failure (NYHA III-IV)
* History of moderate or severe liver failure (Child-Pugh B-C)
* Current or former depression with suicidal ideation
* Topical therapy (anti-inflammatory) for chronic hand eczema 14 days before randomization
* Topical therapy (anti-inflammatory) for chronic hand eczema during study
* Systemic therapy for chronic hand eczema 28 days before randomization
* Systemic therapy for chronic hand eczema during study
* Current treatment with oral dicloxacillin or macrolide
* Current treatment with topical antibiotics
* Diagnosis of contact eczema of clinical significance 3 months before randomization
* Previous treatment with apremilast (Otezla®) or roflumilast (Daxas®)
* Confirmed pregnancy
* Breast feeding
* Blood donation during study
* Allergy to roflumilast or any other PDE-4 inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving at least 75% reduction in hand eczema severity index (HECSI75) at week 16 when compared to HECSI at baseline. | Through study completion, an average of 28 weeks
  HECSI is a measure of hand eczema disease severity considering the extent and intensity of the disease. Each hand is divided into five areas (fingertips, fingers (except the tips), palms, back of hands and wrists) and each area is graded on the intensity of six clinical signs: erythema, induration/papulation, vesicles, fissuring, scaling, and oedema. The grading scale used is: 0, no skin change; 1, mild disease; 2, moderate and 3, severe. The affected area for each location (total of both hands) are given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms. Finally, the total sum of the intensity of the six clinical signs multiplied by the extent of each location is called HECSI score and it may vary from 0 to a maximum of 360 points, with higher scores reflecting greater disease severity. The score reflects HE severity as following: 1-16, mild HE; 17-37, moderate HE; 38-116 severe HE and 117-360, very severe HE.

SECONDARY OUTCOMES:
Proportion of patients achieving at least 50% reduction in baseline HECSI (HECSI50) at assessments. | Through study completion, an average of 28 weeks
  HECSI is a measure of hand eczema disease severity considering the extent and intensity of the disease. Each hand is divided into five areas (fingertips, fingers (except the tips), palms, back of hands and wrists) and each area is graded on the intensity of six clinical signs: erythema, induration/papulation, vesicles, fissuring, scaling, and oedema. The grading scale used is: 0, no skin change; 1, mild disease; 2, moderate and 3, severe. The affected area for each location (total of both hands) are given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms. Finally, the total sum of the intensity of the six clinical signs multiplied by the extent of each location is called HECSI score and it may vary from 0 to a maximum of 360 points, with higher scores reflecting greater disease severity. The score reflects HE severity as following: 1-16, mild HE; 17-37, moderate HE; 38-116 severe HE and 117-360, very severe HE.
Proportion of patients achieving at least 90% reduction in baseline HECSI (HECSI90) at assessments. | Through study completion, an average of 28 weeks
  HECSI is a measure of hand eczema disease severity considering the extent and intensity of the disease. Each hand is divided into five areas (fingertips, fingers (except the tips), palms, back of hands and wrists) and each area is graded on the intensity of six clinical signs: erythema, induration/papulation, vesicles, fissuring, scaling, and oedema. The grading scale used is: 0, no skin change; 1, mild disease; 2, moderate and 3, severe. The affected area for each location (total of both hands) are given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms. Finally, the total sum of the intensity of the six clinical signs multiplied by the extent of each location is called HECSI score and it may vary from 0 to a maximum of 360 points, with higher scores reflecting greater disease severity. The score reflects HE severity as following: 1-16, mild HE; 17-37, moderate HE; 38-116 severe HE and 117-360, very severe HE.
Proportion of patients achieving at least 100% reduction in baseline HECSI (HECSI100) at assessments | Through study completion, an average of 28 weeks
  HECSI is a measure of hand eczema disease severity considering the extent and intensity of the disease. Each hand is divided into five areas (fingertips, fingers (except the tips), palms, back of hands and wrists) and each area is graded on the intensity of six clinical signs: erythema, induration/papulation, vesicles, fissuring, scaling, and oedema. The grading scale used is: 0, no skin change; 1, mild disease; 2, moderate and 3, severe. The affected area for each location (total of both hands) are given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms. Finally, the total sum of the intensity of the six clinical signs multiplied by the extent of each location is called HECSI score and it may vary from 0 to a maximum of 360 points, with higher scores reflecting greater disease severity. The score reflects HE severity as following: 1-16, mild HE; 17-37, moderate HE; 38-116 severe HE and 117-360, very severe HE.
Percent change from baseline in HECSI score at assessments. | Through study completion, an average of 28 weeks
  HECSI is a measure of hand eczema disease severity considering the extent and intensity of the disease. Each hand is divided into five areas (fingertips, fingers (except the tips), palms, back of hands and wrists) and each area is graded on the intensity of six clinical signs: erythema, induration/papulation, vesicles, fissuring, scaling, and oedema. The grading scale used is: 0, no skin change; 1, mild disease; 2, moderate and 3, severe. The affected area for each location (total of both hands) are given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms. Finally, the total sum of the intensity of the six clinical signs multiplied by the extent of each location is called HECSI score and it may vary from 0 to a maximum of 360 points, with higher scores reflecting greater disease severity. The score reflects HE severity as following: 1-16, mild HE; 17-37, moderate HE; 38-116 severe HE and 117-360, very severe HE.
Change (2 or more points) in physician global assessment for chronic hand eczema IGA-CHE) at assessments. | Through study completion, an average of 28 weeks
  The IGA-CHE rates the severity of the patient's global disease assessed by the physician and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Change from baseline in dermatology life quality index (DLQI) at assessments. | Through study completion, an average of 28 weeks
  DLQI is a validated, self-administered, 10-item questionnaire that measure the impact of skin disease on patients' quality of life, based on recall over the past week. Domains include symptoms, feeling, daily activities, social, leisure, work or studying, personal relationships, and treatment. Each question is answered on a scale of 0 (not at all) to 3 (very much) and the total score may vary from 0 to 30.
Change from baseline in patient's global assessment (PaGA) at assessments. | Through study completion, an average of 28 weeks
  The PaGA rates the severity of the patient's global disease assessed by the patient and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Change from baseline in numeric rating scale (NRS) - Peak skin pain on hands within the last 24 hours at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in numeric rating scale (NRS) - Peak skin pain on hands within the last 7 days at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in NRS - Peak itch on hands within the last 24 hours at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in NRS - Peak itch on hands within the last 7 days at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in NRS - sleeplessness within the last 24 hours at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in NRS - sleeplessness within the last 7 at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient symptoms such as pain, itch and sleeplessness on a scale from 0 (no pain, no itch, no sleeplessness) to 10 (worst pain, worst itch, worst sleeplessness).
Change from baseline in NRS - Patient treatment satisfaction within the last 7 at assessments. | Through study completion, an average of 28 weeks
  NRS is a simple and commonly used numeric scale in which the patient rates patient treatment satisfaction on a scale from 0 (very unsatisfied) to 10 (very satisfied).
Change from baseline in quality of life hand eczema questionnaire (QOLHEQ) at assessments. | Through study completion, an average of 28 weeks
  QOLHEQ is a validated, self-administered 30-question questionnaire that measures impairment of health-related quality of life (HRQoL) in patients with HE. Domains include symptoms, emotions, functioning and treatment/prevention. 0 (not at all) to 4 (all the time) and the total score may vary from 0 to 120. A QOLHEQ score greater than 86 is indicative of very strong impairment.
Change from baseline in work productivity and activity impairment: CHE (WPAI:CHE) at assessments. | Through study completion, an average of 28 weeks
  WPAI is a validated, self-administered questionnaire that measures the impact of CHE on work. Domains include time missed from work and impairment of work and regular activities due to CHE.
Adverse events (AEs), serious adverse events (SAEs), serious adverse reactions (SARs), and suspected unexpected serious adverse reactions (SUSARS) documented at assessments. | Through study completion, an average of 28 weeks
  AE are any unfavorable and/or unintended sign or incident, symptoms or disease, whether related to roflumilast or placebo. This also includes laboratory results outside the reference range, though only laboratory results with clinical relevance will be examined. Any AE from the first administration of the trial medication to 8 days after the last administration of the trial medicine will be recorded, though unfavorable event reported in questionnaires will not be recorded as AE. SAE and SAR are any AE or adverse reaction that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a congenital anomaly of birth defect.

OTHER OUTCOMES:
Change in lung function between baseline and week 16 | 16 weeks
  Exploratory outcome: Fractional concentration of exhaled nitric oxide (FeNO) test will be used to evaluate changes in lung function.
  FeNO test will be used to determine the level of eosinophilic lung inflammation. It is performed using a portable device that measures levels of nitric oxide in in parts per billion (PPB) in exhaled air. When the test is performed it is very important that the patient exhales slowly. The test is non-invasive and safe and takes approx. 30 seconds. The test is performed using a NIOX VERO apparatus which is CE-marked.
Change in lung function between baseline and week 16 | 16 weeks
  Exploratory outcome: Spirometry will be used to evaluate changes in lung function.
  Spirometry is the most common pulmonary function test and measures forced expiratory volume during first second (FEV1) and forced volume capacity (FVC). The FEV1/FVC-ratio is used to diagnose obstructive and restrictive lung disease. The test is completed once two acceptable and reproductible measurements have been obtained. The test takes 5-10 minutes and is safe and non-invasive.
Change in natural moisturizing factor (NMF) between baseline and week 16 | 16 weeks
  Exploratory outcome: change in NMF will be assessed using tape-strips.
Change in cytokine levels between baseline and week 16 | 16 weeks
  Exploratory outcome: cytokine analyses by meso scale discovery (MSD) will be done to investigate changes in the epidermal barrier disruption through changes in cytokines (e.g. IL-10).Cytokine levels will be assessed using tape-strips.
Change in ceramides (lipids) between baseline and week 16 | 16 weeks
  Exploratory outcome: lipidomic profiling by high performance liquid chromatography (HP-LC) will be done. Ceramides will be assessed using tape-strips.
Change in skin bacterial communities between baseline and week 16 | 16 weeks
  Exploratory outcome: subsequent microbiome characterization with 16S rRNA sequencing will be done. Changes in the skin microbiome is measured as relative abundance (%) of bacterial genera. Skin microbiome will be assessed using standard eSwaps.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of dermatology and veneorology, Bispebjerg Hospital, Copenhagen, Denmark